CLINICAL TRIAL: NCT03837483
Title: A Single Arm, Open-label Clinical Trial of Hematopoietic Stem Cell Gene Therapy With Cryopreserved Autologous CD34+ Cells Transduced With Lentiviral Vector Encoding WAS cDNA in Subjects With Wiskott-Aldrich Syndrome (WAS)
Brief Title: A Clinical Study to Evaluate the Use of a Cryopreserved Formulation of OTL-103 in Subjects With Wiskott-Aldrich Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione Telethon (Other)
Collaborators: Ospedale San Raffaele (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTL-103-4; 2018-003842-18 (EudraCT Number)
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Wiskott-Aldrich Syndrome
MeSH Terms: conditions — Wiskott-Aldrich Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gene Therapy (Experimental): OTL-103, Autologous CD34+ hematopoietic stem cells transduced ex vivo with a lentiviral vector encoding the human WAS gene
  Interventions: Genetic: OTL-103

INTERVENTIONS:
Genetic: OTL-103 — Autologous hematopoietic stem cells collected from mobilized peripheral blood transduced ex vivo with a lentiviral vector encoding the WAS cDNA

SUMMARY:
This is an open-label, single arm study to evaluate the cryopreserved formulation of OTL-103 Gene Therapy. OTL-103 consists of autologous CD34+ hematopoietic stem cells in which the gene encoding for the Wiskott-Aldrich Syndrome is introduced by means of a third generation lentiviral vector.

ELIGIBILITY:
Inclusion Criteria:

* Age: up to 65 years
* Diagnosis of WAS defined by genetic mutation and at least one of the following criteria:

  * Severe Wiskott-Aldrich Syndrome (WAS) gene mutation, defined by literature data (genotype/phenotype studies).;
  * Absent WASP expression, assessed by flow cytometry;
  * Severe clinical score (Zhu clinical score ≥ 3);
* No human leukocyte antigen (HLA)-identical related donor available for hematopoietic stem cells transplant (HSCT).

Exclusion Criteria:

* End-organ dysfunction, severe active infection not responsive to treatment or other severe disease or clinical condition which, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
* Malignant neoplasia (except local skin cancer) or a documented history of hereditary cancer syndrome.
* Myelodysplasia, cytogenetic alterations characteristic of myelodysplastic syndrome and acute myeloid leukaemia , or other serious haematological disorders
* Documented human immunodeficiency virus (HIV) infection
* Prior allogeneic hematopoietic stem cell transplantation, with evidence of residual cells of donor origin
* Symptomatic herpes zoster, not responsive to specific treatment
* Evidence of acute tuberculosis
* Acute or chronic stable Hepatitis B
* Presence of positive Hepatitis C RNA test result at screening
* Patients not eligible for mobilization protocols in order to obtain CD34+ cells
* Previous Gene Therapy

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-01-21 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of severe infections from 6 to 18 months after gene therapy compared with 1 year before gene therapy | 18 months
Annualized rate of moderate and severe bleeding episodes up to 1 year after gene therapy compared with 1 year before gene therapy | 12 months

SECONDARY OUTCOMES:
Evaluation of the overall survival | 36 months
Number of patients with Vector copy number (VCN)/cell > 0.1 measured in peripheral blood-derived CD3+ cells | 2 years
Percentage of WAS protein expression increased from pre-treatment levels in lymphocytes | 2 years
Percentage of WAS protein expression increased from pre-treatment levels in platelets | 2 years
Number of participants with successful engraftment of OTL-103 | 6 months
  Engraftment of of OTL-103 is measured by hematological reconstitution of an absolute neutrophil count > 500 cell/ul
The number of subjects presenting with malignancies or abnormal clonal proliferation | 2 years

CONTACTS AND LOCATIONS:
Locations (2):
- Children's Healthcare of Atlanta, Inc, Atlanta, Georgia, United States
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Quaranta P, Basso-Ricci L, Jofra Hernandez R, Pacini G, Naldini MM, Barcella M, Seffin L, Pais G, Spinozzi G, Benedicenti F, Pietrasanta C, Cheong JG, Ronchi A, Pugni L, Dionisio F, Monti I, Giannelli S, Darin S, Fraschetta F, Barera G, Ferrua F, Calbi V, Ometti M, Di Micco R, Mosca F, Josefowicz SZ, Montini E, Calabria A, Bernardo ME, Cicalese MP, Gentner B, Merelli I, Aiuti A, Scala S. Circulating hematopoietic stem/progenitor cell subsets contribute to human hematopoietic homeostasis. Blood. 2024 May 9;143(19):1937-1952. doi: 10.1182/blood.2023022666. PMID 38446574